CLINICAL TRIAL: NCT01607372
Title: A Randomized, Double Blind, Placebo-controlled Study to Investigate the Safety and Pharmacodynamics of Repeat Intranasal Administration of the TLR7 Agonist GSK2245035 in Subjects With Respiratory Allergies
Brief Title: A Study to Investigate the Safety and Pharmacodynamics of Repeat Intranasal Administration of the TLR7 Agonist GSK2245035 in Subjects With Respiratory Allergies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 116392
Record Dates: First submitted 2012-03-29; First posted 2012-05-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Asthma and Rhinitis
Keywords: TLR7 agonist, Respiratory Allergies, Allergic Rhinitis, Mild Allergic Asthma, Repeat Dose Safety, Reduction of Allergic Reactivity
MeSH Terms: conditions — Asthma; Rhinitis; Rhinitis, Allergic | interventions — GSK2245035

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK2245035 - 40 ng or placebo (Experimental): Subjects will receive GSK2245035 - 40 nanogram (ng) or placebo once per week for four treatment weeks. There will be washout period of 7 days between treatment periods. GSK medical monitor will review all available clinical and laboratory safety data and decide if subjects can proceed to the next scheduled dosing cohort.
  Interventions: Drug: GSK2245035; Device: Type 1 amber glass bottle; Other: Placebo
- GSK2245035 - 80 ng or placebo (Experimental): Subjects will receive GSK2245035 - 80 ng or placebo once per week for four treatment weeks. There will be washout period of 7 days between treatment periods. GSK medical monitor will review all available clinical and laboratory safety data and decide if subjects can proceed to the next scheduled dosing cohort.
  Interventions: Drug: GSK2245035; Device: Type 1 amber glass bottle; Other: Placebo
- GSK2245035 - 120 ng or placebo (Experimental): Subjects will receive GSK2245035 - 120 ng or placebo once per week for four treatment weeks. There will be washout period of 7 days between treatment periods. GSK medical monitor will review all available clinical and laboratory safety data and decide if subjects can proceed to the next scheduled dosing cohort.
  Interventions: Drug: GSK2245035; Device: Type 1 amber glass bottle; Other: Placebo
- GSK2245035 - 160 ng or placebo (Experimental): Subjects will receive GSK2245035 - 160 ng or placebo once per week, for four treatment weeks. There will be washout period of 7 days between treatment periods.
  Interventions: Drug: GSK2245035; Device: Type 1 amber glass bottle; Other: Placebo

INTERVENTIONS:
Drug: GSK2245035 — GSK2245035 nasal spray solution. A solution formulation in saline, preserved with Benzalkonium Chloride and Disodium Edetate
Device: Type 1 amber glass bottle — fitted with a metered Valios VP7 pump
Other: Placebo — As for GSK2245035 nasal spray solution except for omission of the active ingredient

SUMMARY:
GSK2245035 is a highly selective Toll-like receptor 7 (TLR7) agonist that stimulates preferentially the induction of type I interferons. Intranasal (i.n.) administration of GSK2245035 in humans causes immune changes in the upper airways milieu that may alter bystander immune responsiveness to aeroallergens and contribute to reduction of allergic reactivity in subjects with respiratory allergies. The purpose of this study is to examine the safety and pharmacodynamics (PD) of repeat dosing with i.n. GSK2245035 in subjects with respiratory allergies. The safety and pharmacodynamic response of four weekly administrations of escalating doses of i.n. GSK2245035 will be investigated and the maximum tolerated dose will be established. The study will be conducted in patients with symptomatic allergic rhinitis and mild asthma. The overall duration of the study will be up to a maximum of approximately 122 days considering 90 days screening period, 22 days treatment period and 10 days follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Good general health, as determined by a responsible and experienced physician, based on a medical evaluation, including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Males between 18 and 62 years of age inclusive.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until four days after the last dosing.
* Females between 18 and 62 years of age inclusive, if they are of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy, or postmenopausal, defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Body weight greater than and equal to 50 kilogram (kg) and body mass index (BMI) within the range 19 - 35 kg/meter square (m^2) (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete all required study measurements.
* Documented history of Symptomatic perennial allergic rhinitis and mild asthma driven by house dust mite (HDM) for more than 3 years, that does not require regular use of inhaled steroids. Subjects with symptomatic perennial allergic rhinitis and mild asthma driven by house dust mite (HDM) will need to have a positive skin allergy test (wheal ≥ 3 millimeter [mm]) or RAST (≥ class 2) to house dust mite allergens. (However, an allergen radio allergosorbent test [RAST] or skin test can be omitted if a subject provides clear evidence confirmed by a physician of an analogous positive test within the last 3 years).

Exclusion Criteria:

* History of immunological disorders or other diseases (including, but not limited to, malignancy, cardiovascular, gastro-intestinal, hepatic, renal, haematological, neurological, endocrine or pulmonary disease) that in the opinion of the investigator and GSK medical monitor may pose additional risk factors
* Nasal conditions that according to the opinion of the investigator may affect the outcome of the study, i.e. nasal septal perforation, nasal polyps, other nasal malformations or history of frequent nosebleeds.
* Respiratory tract infection within 4 weeks prior to the first dosing.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody
* A positive screening or pre-dose drug/alcohol screen
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 14 drinks for males or greater than 7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 millileter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Participation in a clinical trial with receipt of an investigational product within 3 months prior to the first dosing day.
* Exposure to more than four new chemical entities within 6 months prior to the first dosing day.
* History of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates participation in this study.
* Donation of blood or blood products in excess of 500 mL within a 56-day period.
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of severe asthma
* Serious asthma exacerbation requiring hospital visit and/ or treatment with oral steroids or high doses of inhaled steroids within 6 weeks prior to screening
* History of treatment with allergen-specific immunotherapy
* Pre-bronchodilator FEV1 less than and equal to 70% of predicted at screening
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to first dosing, unless in the opinion of the investigator and GlaxoSmithKline (GSK) medical monitor the medication will not interfere with the study procedures or compromise subject safety. Paracetamol is an exception and will be permitted at daily doses of up to 4 g from screening to follow-up. During the dosing visits Paracetamol can be used, if needed, only if the investigator allows it.
* Subjects using steroid treatment for allergic rhinitis and/or asthma may participate in the study if they can remain free of medication throughout the study period starting from the following periods of time prior to first dosing: Nasal steroids: 4 weeks; Oral steroids: 12 weeks; Inhaled steroids: 4 weeks
* Subjects using other medications for their allergic rhinitis and/or asthma on an as needed basis may participate in the study if they can abstain from: Xanthines (including theophylline, but not including caffeine), anticholinergics, cromoglycates, leukotriene antagonists, 5-lipoxygenase inhibitors and longacting inhaled beta-agonists from 1 week prior to screening and throughout the study Na; Nasal antihistamines: 48 hours prior each dosing; Oral antihistamines: 76 hours prior each dosing; Nasal decongestants: 24 hours prior each dosing; Oral decongestants: 24 hours prior each dosing; Short acting inhaled beta-agonists: 48 hours prior each dosing

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing adverse events (AEs) | Up to 122 Days
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Hematology parameters as a safety measure | Up to 112 Days
  The hematology parameters included are platelet count, red blood cell (RBC) count, white blood cell (WBC) count, reticulocyte count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), neutrophils, lymphocytes, monocytes, eosinophils, basophils.
Clinical Chemistry parameters as a safety measure | Up to 112 Days
  Clinical chemistry parameters included are blood urea nitrogen (BUN), creatinine, glucose, potassium, C-Reactive protein (CRP) potassium, chloride, total carbon dioxide, calcium, total and direct bilirubin, Aspartate transaminase (AST), Alanine transaminase (ALT), alkaline phosphatase, uric acid, protein and albumin
Urinalysis parameters as a safety measure | Up to 112 Days
  Urinalysis parameters included are specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick, microscopic examination (if blood or protein is abnormal)
Body temperature | Up to 112 Days
Systolic and diastolic blood pressure (BP) | Up to 112 Days
Pulse rate | Up to 112 Days
ECG parameters | Up to 112 Days
  A 12 lead electrocardiogram (ECG) will be measured using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Nasal examination | Up to 112 Days
  Visual nasal examination will be conducted by a trained physician
Nasal symptoms assessment | Up to 23 Days
  Nasal tolerability symptoms itching, discomfort, post-nasal drip, rhinorrhoea, obstruction will be assessed using a Visual analogue score system

SECONDARY OUTCOMES:
FEV1 assessment | Up to 112 Days
  To evaluate the effect of four repeat doses of i.n. GSK2245035 administered once per week on lung function, as measured by Forced expiratory volume in one second FEV1
TLR7-induced blood PD biomarkers, including TLR7-induced cytokines | Up to 23 Days
  To evaluate the induction of TLR7-associated blood PD biomarkers following administration of i.n. GSK2245035 once per week
TLR7-induced nasal PD biomarkers, including but not limited to induced protein (IP)-10, i.n. nasal lavage fluid | Up to 23 Days
  To evaluate the induction of TLR7-associated nasal PD biomarkers following administration of repeat doses of i.n. GSK2245035 once per week
Daily rhinitis symptoms and use of medication diaries during the study period | Up to 122 Days
Daily asthma symptoms and use of medication diaries during the study period | Up to 122 Days
Daily morning peak expiratory flow (PEF) during the study period | Up to 112 Days
Exhaled NO assessment | Up to 23 Days
Cell counts and differential in nasal lavage | Up to 23 Days
Exploratory allergic biomarkers including but not limited to immunoglobulins and cytokines in blood and nasal lavage fluid and tissue | Up to 23 Days
Plasma GSK2245035 concentrations | Up to 23 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tsitoura D, Ambery C, Price M, Powley W, Garthside S, Biggadike K, Quint D. Early clinical evaluation of the intranasal TLR7 agonist GSK2245035: Use of translational biomarkers to guide dosing and confirm target engagement. Clin Pharmacol Ther. 2015 Oct;98(4):369-80. doi: 10.1002/cpt.157. PMID 26044169
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116392 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register